CLINICAL TRIAL: NCT02037204
Title: Instant MSC Product Accompanying Autologous Chondron Transplantation (IMPACT): Safety and Feasibility of a Single-stage Procedure for Focal Cartilage Lesions of the Knee.
Brief Title: IMPACT: Safety and Feasibility of a Single-stage Procedure for Focal Cartilage Lesions of the Knee.
Acronym: IMPACT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, D.B.F. Saris, MD, PhD, Orthopaedic surgeon, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMPACT
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Results first posted 2019-01-02 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-06

CONDITIONS: Foreign-Body Reaction; Inflammation; Effusion (L) Knee; Knee Pain Swelling
Keywords: IMPACT; Chondrons; Mesenchymal stem cells; Allogeneic MSCs; single-stage; Cartilage repair; Safety; Efficacy
MeSH Terms: conditions — Foreign-Body Reaction; Inflammation; Tooth, Impacted

STUDY DESIGN:
Intervention Model Description: First in man surgery: autologous chondrons are mixed with allogeneic MSCs and implanted in a fibrin glue carrier in a one-stage surgical procedure.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cartilage repair surgery (Experimental): Single-stage cartilage repair surgery using autologous chondrons (10-20%) and allogeneic MSCs (80-90%) in a fibrin glue carrier with a dosage of two million cells/ cm2 applied once during a surgical procedure.
  Interventions: Other: Cartilage repair surgery

INTERVENTIONS:
Other: Cartilage repair surgery — Single-stage surgery, After debridement, the cartilage defect is filled with the fibrin glue carrier containing autologous chondrons and allogeneic MSCs
  Other Names: Single-stage; Cartilage repair; IMPACT

SUMMARY:
Articular cartilage defects in the knee have a poor intrinsic healing capacity and may lead to functional disability and osteoarthritis. Cartilage cell therapy using autologous chondrocyte implantation (ACI) has been established as the first advanced treatment therapy medicinal product. Although this technique has achieved good mid-term results, it is a costly and extensive two-stage procedure which is limited by the number of chondrocytes obtained by biopsy and the dedifferentiation resulting from the expansion phase. Therefore, there is a need for improvement. A new cartilage repair technique should aim at decreasing surgical trauma, lowering complexity, improving logistics and cost-effectiveness while retaining or improving clinical outcome. Direct contact between mesenchymal stromal cells (MSCs) and dedifferentiated articular chondrocytes in vitro showed improvement of the chondrogenic phenotype of dedifferentiated articular chondrocytes. In addition, preserving the pericellular matrix of chondrocytes improves cartilage formation. These chondrons (chondrocytes with their pericellular matrix) have shown improved cartilage formation when combined with allogeneic MSCs in extensive preclinical studies. The cells are mixed with fibrin cell carrier and applied to the cartilage lesion within one surgical procedure. This will reduce patient morbidity and improve patient care through immediate transplantation of a potent cell-based cartilage product. This is a phase I/II prospective monocenter study to evaluate the safety and feasibility of the IMPACT for treatment of focal articular cartilage lesions of the knee.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 and <45 years old
* Symptomatic isolated full-thickness articular cartilage lesion on the femoral condyle or trochlea.
* Size 2 - 8 cm2
* Intact anterior cruciate ligament

Exclusion Criteria:

* (History of) osteoarthritis, defined as Kellgren-Lawrence grade >3 as determined from appropriate X-ray.
* Concomitant inflammatory disease that affects the joint (rheumatoid arthritis, metabolic bone disease, psoriasis, gout, symptomatic chondrocalcinosis)
* (History of) Septic arthritis.
* Malalignment requiring an osteotomy.
* (History of) total menisectomy in the target knee joint.
* Any surgery in the knee joint 6 months prior to study inclusion.
* Risk groups for MRI scanning due to the magnetic field like patients with pacemakers, nerve stimulators, metal particles, stents, clips or implants, (possible) pregnancy or breast feeding.
* Patients with severe anxiety for MRI scans and/or needles

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2013-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tommy S. de Windt, MD, Study Director — UMC Utrecht; Daniel B.F. Saris, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

REFERENCES:
- [Background] Bekkers JE, Creemers LB, Tsuchida AI, van Rijen MH, Custers RJ, Dhert WJ, Saris DB. One-stage focal cartilage defect treatment with bone marrow mononuclear cells and chondrocytes leads to better macroscopic cartilage regeneration compared to microfracture in goats. Osteoarthritis Cartilage. 2013 Jul;21(7):950-6. doi: 10.1016/j.joca.2013.03.015. Epub 2013 Apr 9. PMID 23583464
- [Background] Bekkers JE, Tsuchida AI, van Rijen MH, Vonk LA, Dhert WJ, Creemers LB, Saris DB. Single-stage cell-based cartilage regeneration using a combination of chondrons and mesenchymal stromal cells: comparison with microfracture. Am J Sports Med. 2013 Sep;41(9):2158-66. doi: 10.1177/0363546513494181. Epub 2013 Jul 5. PMID 23831891
- [Background] Vonk LA, Doulabi BZ, Huang C, Helder MN, Everts V, Bank RA. Preservation of the chondrocyte's pericellular matrix improves cell-induced cartilage formation. J Cell Biochem. 2010 May;110(1):260-71. doi: 10.1002/jcb.22533. PMID 20213765
- See also: Trials Register of the European Union — https://www.clinicaltrialsregister.eu/ctr-search/trial/2012-001570-29/NL
- See also: IMPACT animation — https://www.youtube.com/watch?v=S3rIBjA03AA

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment started on February 1st 2013 and was completed in September 2014
Pre-assignment Details: Four patients were excluded based on MRI scans showing multiple cartilage defects and/ or osteochondral defects. Inclusion was continued until n = 35 was reached
Groups:
- Cartilage Repair Surgery: All 35 patients received a single-stage cartilage repair treatment using autologous chondrons and allogeneic MSCs in a fibrin glue carrier.
Period: Overall Study
Arm/Group | Cartilage Repair Surgery
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Cartilage Repair Surgery: Single-stage cartilage repair surgery using autologous chondrons and allogeneic MSCs in a fibrin glue carrier.
  Cartilage repair surgery: Single-stage surgery, After debridement, the cartilage defect is filled with the fibrin glue carrier containing autologous chondrons and allogeneic MSCs
Arm/Group | Cartilage Repair Surgery
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 24
Region of Enrollment [Number; unit: participants]
  Netherlands | 35

OUTCOME MEASURES:

1. Primary Outcome: Safety: Adverse Events
Description: Adverse events rate
Time Frame: 18 months
Population: All patients were monitored for the duration of the studie for inflammation and signs of a foreign body response by an independent physician using standardized clinical measures, pain assessment by numeric rating scale for pain and blood analysis including serum C-reactive protein, erythrocyte sedimentation rate and leukocyte count.
Measure: Number; unit: participants
Groups:
- Cartilage Repair Surgery: Single-stage cartilage repair surgery in 35 patients, using autologous chondrons and allogeneic MSCs in a fibrin glue carrier.
Arm/Group | Cartilage Repair Surgery
Number analyzed (Participants) | 35
participants | 0

2. Secondary Outcome: Clinical Improvement, Knee Injury and Osteoarthritis Outcome Score
Description: Clinical improvement as measured by patient reported outcome scores. The questionnaire has been developed to evaluate the symptoms and limitations for patients with osteoarthritis. The outcome of the KOOS-scale varies from 0-100, where 0 indicates the greatest possible problems and is the worst outcome and 100 indicates no problems.
Time Frame: 3 and 18 months
Population: Differences in clinical outcome between baseline and 3 and 12 months after surgery were tested by a repeated measures analysis of variance (ANOVA).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Cartilage Repair Surgery: To evaluate the clinical status of the patients treated with the IMPACT therapy, the included patients were asked to complete the Knee injury and Osteoarthritis Outcome Scoring (KOOS), The visual analog scale (VAS) for pain and the EuroQoL 5-Dimension Health Questionnaire (EQ5D) at baseline (before IMPACT therapy) and at 3, 6, and 12 months follow-up.
Arm/Group | Cartilage Repair Surgery
Number analyzed (Participants) | 35
units on a scale
  KOOS outcome baseline | 57.9 (16.1)
  KOOS outcome 3 months | 76.6 (11.1)
  KOOS outcome 18 months | 85.4 (13.3)
Statistical Analysis 1: Comparison: Cartilage Repair Surgery; A repeated-measures analysis of variance was used to test for differences in clinical outcome between baseline and 3, and 18 months after surgery; Test type: Non-Inferiority — A repeated-measures analysis of variance was used to test for differences in clinical outcome between baseline and 3, and 18 months after surgery; p < 0.05, ANOVA

3. Other Pre Specified Outcome: Structural Repair
Description: To examine parameters of structural repair at one year after treatment using MRI and a second-look arthroscopy.
Time Frame: 12 months
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Health Care Use and Costs
Description: To assess the healthcare use and costs related to the procedure as well as the health-related work leave during the study period.
Time Frame: 18 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All patients were monitored for the duration of 18 months after surgery, at fixed time points (at 7 days, 6 weeks and 3,6,12 and 18 months after surgery), for inflammation and signs of a foreign body response by an independent physician (rheumatologist) using standardized clinical measures, pain assessment by numeric rating scale for pain and blood analysis including serum C-reactive protein (CRP), erythrocyte sedimentation rate (ESR) and leukocyte count.
Arm/Group | Cartilage Repair Surgery
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 18/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cartilage Repair Surgery (N=35)
Post surgery (joint swelling, pain) (Musculoskeletal and connective tissue disorders) | 18 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No